CLINICAL TRIAL: NCT02579421
Title: Sex Differences and Progesterone: Association With Impulsivity and Marijuana Reduction in Co-Users of Marijuana and Nicotine Cigarettes
Brief Title: Hormones and Reduction in Co-users of Marijuana and Nicotine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015NTLS141
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Marijuana Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Progesterone; Crinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Males - Progesterone (Active Comparator): 200 mg progesterone BID
  Interventions: Drug: Progesterone
- Males - Placebo (Placebo Comparator): placebo BID
  Interventions: Drug: placebo
- Females - Progesterone (Active Comparator): 200 mg progesterone BID
  Interventions: Drug: Progesterone
- Females - Placebo (Placebo Comparator): placebo BID
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Progesterone — generic progesterone
  Other Names: Promitrium, Crinone, Endometrin, Prochieve
  Arms: Females - Progesterone; Males - Progesterone
Drug: placebo — placebo
  Arms: Females - Placebo; Males - Placebo

SUMMARY:
The purpose of this study is to examine the role of progesterone (a naturally occurring hormone found in both men and women) on reducing marijuana use. The investigators will see if progesterone effects impulsivity, withdrawal, mood and stress during marijuana cessation.

DETAILED DESCRIPTION:
This double-blind, randomized pilot clinical trial will prescreen an estimated 250 potential subjects, consent and further evaluate approximately 100 potential subjects, and ultimately enroll 70 subjects to ensure 40 subjects will provide a primary marijuana reduction outcome measure at four weeks post quit date. Subjects will be stratified by sex then randomized to one of two treatment groups (n=20 per drug group, 50% female): progesterone (PRO; 200mg 2x/day) or Placebo (PBO). Telephone screening and visit invitation (20 minutes) leads to the consent process and in-person screening including medical-psychiatric evaluation for inclusion/exclusion (two visits, two hours each), then randomization and medication start (7 days), then stable medication (28 days) with medication reduction and final evaluation (7 days).

ELIGIBILITY:
Inclusion Criteria:

* Males 18-60 years old, females 18-50 years old
* Stable physical and mental health
* Self-report Timeline Follow-Back (TLFB) indicating current marijuana use ≥4 days/week for ≥1 year
* Positive urine THC dipstick test (> 50ng/mL; indicating marijuana use in the past 48-72 hours)
* Motivated to change their marijuana use (>1 on a 10-point Likert-type scale) -Regular or sporadic use of nicotine cigarettes (> 1 cigarettes in the past 30 days) -Self-report of regular menstrual cycles >6 months (female only)
* Willing to use double-barrier contraception if sexually active and not surgically sterilized (female only)
* Ability to comply with study procedures, ability to provide informed consent.

Exclusion Criteria:

* Current breastfeeding (females only),
* Current or planned pregnancy within the next three months (females only)
* DSM-IV diagnoses for psychotic disorders, bipolar disorder, ADHD, major depressive disorder within the last 3 months
* Substance dependence within the last 3 months with the exception of nicotine and marijuana dependence
* Unstable psychotropic medications (<3 months)
* Current use of exogenous hormones, finasteroid (propecia), efavirenz, red clover, ketoconazole and other drugs that are CYP3A4 inhibitors
* Conditions contraindicated to progesterone treatment (including, but not limited to, thrombophlebitis, deep vein thrombosis, pulmonary embolus, clotting or bleeding disorders, heart disease, diabetes, history of stroke, allergy to peanuts, hypersensitive to progesterone and liver dysfunction)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Allen, Ph.D,M.D., Principal Investigator — University of Minnesota
Locations (1):
- Delaware Clinical Research Unit, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone - Males: 200 mg progesterone BID
  Progesterone: generic progesterone
- Placebo - Males: placebo BID
  placebo: placebo
- Progesterone - Females: 200 mg progesterone BID
- Placebo - Females: pacebo BID
Period: Overall Study
Arm/Group | Progesterone - Males | Placebo - Males | Progesterone - Females | Placebo - Females
Started | 23 | 23 | 6 | 6
Completed | 17 | 18 | 5 | 3
Not Completed | 6 | 5 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Progesterone - Females: 200 mg progesterone BID
  Progesterone: generic progesterone
- Placebo - Females: placebo BID
  placebo: placebo
- Total: Total of all reporting groups
Arm/Group | Progesterone - Males | Placebo - Males | Progesterone - Females | Placebo - Females | Total
Number analyzed (Participants) | 23 | 23 | 6 | 6 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (11.3) | 40.7 (10.9) | 34.0 (7.7) | 37.0 (7.6) | 38.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 6 | 6 | 12
  Male | 23 | 23 | 0 | 0 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 9 | 1 | 1 | 18
  White | 13 | 12 | 2 | 2 | 29
  More than one race | 3 | 1 | 2 | 2 | 8
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 6 | 6 | 58
Baseline MJ use per day [Mean (Standard Deviation); unit: MJ use occasions per day] | 14.7 (6.2) | 13.9 (8.6) | 12.6 (8.6) | 12.0 (4.4) | 14.7 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Marijuana Use as Defined by the TLFB
Description: Marijuana use as defined by the TLFB at the week 4 visit relative to the baseline visit.
Time Frame: 5 weeks. Baseline to week 4
Population: Some participant data was not included in the analysis because it was missing
Measure: Mean (Standard Deviation); unit: MJ use occasions per day
Arm/Group | Males - Progesterone | Males - Placebo | Females - Progesterone | Females - Placebo
Number analyzed (Participants) | 17 | 18 | 5 | 3
MJ use occasions per day | -1.7 (0.8) | -1.4 (1.1) | -0.9 (1.0) | -2.9 (1.0)

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Progesterone - Males | Placebo - Males | Progesterone - Females | Placebo - Females
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT02579421/Prot_SAP_000.pdf